CLINICAL TRIAL: NCT05204550
Title: A Randomised, Placebo-controlled Trial to Investigate the Efficacy of Intranasal Heparin Treatment to Reduce Transmission of SARS-CoV-2 Infection and COVID 19 Disease Among Household Contacts of SARS-CoV-2+ Adults and Children
Brief Title: Intranasal Heparin Treatment to Reduce Transmission Among Household Contacts of COVID 19 Positive Adults and Children
Acronym: INHERIT
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Murdoch Childrens Research Institute (Other)
Collaborators: University of Melbourne (Other); Northern Hospital, Australia (Other); Monash University (Other); The Peter Doherty Institute for Infection and Immunity (Other); St Vincent's Hospital Melbourne (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 83609
Record Dates: First submitted 2022-01-21; First posted 2022-01-24 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Heparin; Sodium Chloride; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- intranasal heparin (Experimental): Unfractionated heparin (UFH) 1400u each nostril (as heparin solution 5,000u/ml, 140 microL/actuation, Two actuations each nostril) Three times daily via a plastic nasal inhalator device (APTAR, UK) for 10 days.
  This is a maximal dose per day of UFH of 8400u. ie 700 x 2 actuations per nostril (1400 x2) 3 times per day (1400x2x3 = 8400u)
  Interventions: Drug: unfractionated heparin
- intranasal saline (Placebo Comparator): Comparator 0.9% saline (as saline solution, 140 microlitres/actuation, Two actuations each nostril) Three times daily via a plastic nasal inhalator device(APTAR, UK) for 10 days.
  Interventions: Drug: 0.9%sodium chloride

INTERVENTIONS:
Drug: unfractionated heparin — intranasal
  Other Names: heparin
  Arms: intranasal heparin
Drug: 0.9%sodium chloride — intranasal
  Other Names: normal saline
  Arms: intranasal saline

SUMMARY:
Coronavirus-induced disease 2019 (COVID-19) is an infection caused by a virus whose full name is severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). This is a new and rapidly-spreading infectious disease which carries a significant risk of death, has brought massive economic impact globally and has proved hard to contain through public health measures. While we currently have effective vaccines, they do not protect the whole community and the constant threat of new mutations means there is an urgent need to identify new approaches to reducing community spread of infection.

Heparin is a naturally occurring sugar molecule which has been used for a century to treat a range of medical problems including heart attacks, strokes, and blood clots. It has also been investigated as a treatment for pneumonias. Recent research suggests it binds to the SARS-CoV-2 virus in such a way it may reduce the virus' ability to enter cells. This may be an important way to tackle the early stages of infection which occurs inside the nose. Therefore, this medication could be used amongst people with early COVID-19 infection and amongst their household contacts to reduce the rate of virus transmission during local outbreaks. If proven effective there are many other potential uses as primary prophylaxis for people working in high risk areas, for travel, for protection in high risk crowded environments such as nightclubs, or sporting events. Heparin is safe, inexpensive, available worldwide and if effective could be rapidly used across the world to slow progression of the current pandemic.

Further there are recent studies suggesting that the risk of brain complications as part of "long COVID", are directly related to the amount of virus in the nose. Reducing the viral load in the nose is thought to be effective in reducing these "long COVID" complications. This study will explore the effect of the intervention on viral load and long COVID.

In this study, researchers want to investigate this medicine in people who have been identified by a COVID-19 swab test to be in the early stages of infection(defined as the index case), and amongst their household contacts. Each participant would take the medicine or a dummy control solution by spray into their nose three times a day for 10 days. The study will investigate if there are fewer people who contract SARS-CoV-2 infection by day 10 amongst households who receive the medicine than households which receive the dummy control.

DETAILED DESCRIPTION:
Multi-centre, prospective, randomised, placebo-controlled two-arm cluster randomised superiority clinical trial.

Individual households with at least one person with Polymerase chain reaction assay(PCR) or Rapid Antigen test (RAT) confirmed SARS-CoV-2 infection will be randomised so that all consenting people in that household receive intranasal heparin or placebo.

The rate of subsequent PCR confirmed SARS-CoV-2 infections in exposed households will be measured to determine the effect of intranasal heparin on reducing transmission to close contacts.

The rate of symptom development in all participants will be used to determine effect of treatment in preventing symptomatic disease The rate of hospitalisation of all participants will be measured to determine the effect of treatment on development of severe disease.

The presence of clinical neurological long COVID symptoms will be assessed at 6 and 12 months to determine the effect of treatment on long COVID.

Objectives Primary

• To test the efficacy of early treatment and post exposure prophylaxis to reduce transmission to household contacts on SARS-CoV-2 PCR assay by day 10.

Secondary

* To test the efficacy of intranasal heparin to reduce SARS-CoV-2 viral shedding: over 10 days from day of positive swab (health professional collected nasopharyngeal swab Day 3 and 5, and Day 10: self-administered anterior nasal swab swab days 1,2,3,4,5 and 10).
* To test the safety of intranasal heparin for treatment of adult and children outpatients with SARS CoV-2 infection
* To test whether intranasal heparin administration reduces symptomatic disease in index cases and household contacts
* To test the impact of intranasal heparin on peak severity of illness.
* Quantification of replication-competent virus.
* To assess the impact of intranasal heparin on long COVID neurological symptoms

ELIGIBILITY:
Inclusion Criteria:

* Any person > 5 years of age who tests positive to SARS-CoV-2 or is a household contact of someone of any age who tests positive is eligible for the trial.
* Index case must be within 72 hours of positive test.
* The positive test can be a RAT or a standard PCR nasal swab performed at an accredited laboratory for the diagnosis of COVID-19 as per the department of health regulations. If initial test is a RAT, then a a standard PCR nasal swab performed at an accredited laboratory for the diagnosis of COVID-19 as per the department of health regulations will be collected prior to randomisation but does not delay entry into the study awaiting the confirmatory result.
* All participants must provide a signed and dated consent form and for children < 16 years have a legally acceptable representative capable of understanding the informed consent document and providing consent on the participant's behalf. Consent forms will be developed in multiple languages and provided in a language that the participants are fluent in speaking.
* At least one other person other than the index case in each household must consent to participation to enable the consenting members of the household to be randomised. Household members who do not consent to participate in the randomised trial but whom consent to have their COVID-19 status recorded can contribute to outcome measures where relevant.

Exclusion Criteria:

Children Age < 5 years are excluded from being randomised to therapy but can contribute to the outcome measures if they are swab negative on day 1.

* Documented Heparin allergy
* Previous documented heparin induced thrombocytopenia (HIT)
* Recurrent epistaxis that has required hospitalisation in last 3 months
* >72 hours since index case tested positive
* Inability to provide patient information and consent forms or study instructions in a language in which the patient is competent.
* Household members who are swab positive on day 1 are excluded from contributing to the primary outcome, but are randomised and still contribute to secondary outcomes

Ages: 5 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 506 (Actual)
Dates: Start 2023-01-30 (Actual); Primary Completion 2024-12-09 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Number of household contacts (swab negative on day 1) testing positive for SARS-CoV-2 by PCR on either of three routine nasopharyngeal swabs on day 3,5 and 10 after enrolment or on nasopharyngeal swab in response to clinical symptoms in the first 14 days | 14 days from randomisation
  household contacts who become COVID 19 positive at any time during study period

SECONDARY OUTCOMES:
Number of household contacts (swab negative on day 1 of study) becoming symptomatic of COVID-19 in next 28 days | 28 days from randomisation
  household contacts who develop symptomatic COVID 19 defined as : fever (≥38°C) PLUS ≥1 respiratory symptom (sore throat, cough, shortness of breath); OR 2 respiratory symptoms (sore throat, cough, shortness of breath); OR 1 respiratory symptom (sore throat, cough, shortness of breath) PLUS ≥2 non-respiratory symptoms (chills, nausea, vomiting, diarrhea, headache, conjunctivitis, myalgia, arthralgia, loss of taste or smell, fatigue or general malaise).
total number of index cases and household contacts (nasopharyngeal swab positive on day 1) combined, who remain swab positive on day 3 | 3 days from randomisation
  proportion of COVID 19 positive participants becoming swab negative by day 3
total number of index cases and household contacts (nasopharyngeal swab positive on day 1) combined, who remain swab positive on day 5 | 5 days from randomisation
  proportion of COVID 19 positive participants becoming swab negative by day 5
total number of index cases and household contacts (nasopharyngeal swab positive on day 1) combined, who remain swab positive on day 10 | 10 days from randomisation
  proportion of COVID 19 positive participants becoming swab negative by day 10
Time to swab negative based on daily anterior nasal swab for index cases and household contacts combined who were swab positive on day 1. | 10 days from randomisation
  mean time to swab negative in all COVID 19 positive participants
Quantitative replication sub genomic viral RNA at days 3 post randomisation. | 3 days from randomisation
  The quantitative assay to generate these data will be the Q2 SARS-CoV-2 Viral Load Quantitation Assay, with lower limit of quantification of 500 copies/ml and upper limit of quantification of 500,000,000 copies/ml. Results below or above these limits will be included in the mean and the mean change from baseline, with imputed value 499 and 500,000,001, respectively. High viral load is defined as >106 copies/mL, low viral load is defined as ≤106 copies/mL, and undetectable viral load is defined as < 500 copies/ml
Quantitative replication sub genomic viral RNA at days 5 post randomisation. | 5 days from randomisation
  The quantitative assay to generate these data will be the Q2 SARS-CoV-2 Viral Load Quantitation Assay, with lower limit of quantification of 500 copies/ml and upper limit of quantification of 500,000,000 copies/ml. Results below or above these limits will be included in the mean and the mean change from baseline, with imputed value 499 and 500,000,001, respectively. High viral load is defined as >106 copies/mL, low viral load is defined as ≤106 copies/mL, and undetectable viral load is defined as < 500 copies/ml
Quantitative replication sub genomic viral RNA at days 10 post randomisation. | 10 days from randomisation
  The quantitative assay to generate these data will be the Q2 SARS-CoV-2 Viral Load Quantitation Assay, with lower limit of quantification of 500 copies/ml and upper limit of quantification of 500,000,000 copies/ml. Results below or above these limits will be included in the mean and the mean change from baseline, with imputed value 499 and 500,000,001, respectively. High viral load is defined as >106 copies/mL, low viral load is defined as ≤106 copies/mL, and undetectable viral load is defined as < 500 copies/ml
The number of participants who discontinue treatment prior to day 10 from randomisation | 10 days from randomisation
  treatment tolerability
Number of index cases and household contacts swab positive on day 1, hospitalized with COVID-19 by day 28 from randomization | 28 days from randomisation
  symptomatic progression of COVID 19
Number of household contacts swab negative on day 1, hospitalized with COVID-19 by day 28 from randomization | 28 days from randomisation
  symptomatic progression of COVID 19
Maximum severity score of participants (index case and household contacts swab positive on day 1 compared to household contacts swab negative on day 1) during the study period as recorded by daily symptom diary up to day 28 | 28 days from randomisation
  A COVID-19 Composite Subjective Symptom Severity Score will be generated using the 11 common symptoms for COVID 19 infection listed at the Center for disease control website and a self-rated symptom severity assessment generated for each symptom on a daily basis using a Likert scale for each symptom (Scale 0-3: not present mild, moderate, severe).
  Common symptoms:
  * Fever or chills
  * Cough
  * Shortness of breath or difficulty breathing
  * Fatigue
  * Muscle or body aches
  * Headache
  * New loss of taste or smell
  * Sore throat
  * Congestion or runny nose
  * Nausea or vomiting
  * Diarrhea
  Index cases and household contacts will be asked to complete symptom severity checklists daily.
  Analysis will utilise a summative score
time to symptom resolution analysis for index case and household contacts swab positive on day 1 compared to household contacts swab negative on day 1, during the study period as measured with daily symptom diary until on day 28 | 28 days from randomisation
  hazard ratio of time to sustained improvement or resolution of symptoms based on daily symptoms reports up to day 28 specific to the 11 common symptoms for COVID 19 infection listed at the Center for Disease Control website and a self-rated symptom severity assessment generated for each symptom on a daily basis using a Likert scale for each symptom (Scale 0-3: not present mild, moderate, severe).
  Common symptoms:
  * Fever or chills
  * Cough
  * Shortness of breath or difficulty breathing
  * Fatigue
  * Muscle or body aches
  * Headache
  * New loss of taste or smell
  * Sore throat
  * Congestion or runny nose
  * Nausea or vomiting
  * Diarrhea
  Index cases and household contacts will be asked to complete symptom severity checklists daily.
Number of participants with clinical symptoms of neurological long COVID at 6 months post initial positive COVID-19 test. | 6 months from randomisation
  Telehealth self-rated symptom assessment using a Likert scale(0-3: absent, mild, moderate, severe). for each symptom Symptoms screened: fatigue, malaise, daytime tiredness, impaired concentration, brain fog, sleep disturbance, forgetfulness, confusion, Headache, dizziness, nausea, Hypo/anosmia , hypo/ageusia, Impaired walking, tingling feet or hands, burning feet or hands, numb feet or hands, impaired fine motor skills, muscle pain, Epilepsy, anxiety, depression. Cognition and mood will be assessed using the harmonised procedures developed by the Neuro-COVID Neuropsychology International Task force. Telephone - Montreal Cognitive Assessment,Patient's Assessment of Own Functioning, Wechsler Adult Intelligence Scale, Digit Span (Forward and Backward),Brief Visuospatial Memory Test - Revised,Hopkins Verbal Learning Test, Depression, Anxiety, Stress Scales
Number of participants with clinical symptoms of neurological long COVID at 12 months post initial positive COVID-19 test. | 12 months from randomisation
  Telehealth self-rated symptom assessment using a Likert scale(0-3: absent, mild, moderate, severe). for each symptom Symptoms screened: fatigue, malaise, daytime tiredness, impaired concentration, brain fog, sleep disturbance, forgetfulness, confusion, Headache, dizziness, nausea, Hypo/anosmia , hypo/ageusia, Impaired walking, tingling feet or hands, burning feet or hands, numb feet or hands, impaired fine motor skills, muscle pain, Epilepsy, anxiety, depression. Cognition and mood will be assessed using the harmonised procedures developed by the Neuro-COVID Neuropsychology International Task force. Telephone - Montreal Cognitive Assessment,Patient's Assessment of Own Functioning, Wechsler Adult Intelligence Scale, Digit Span (Forward and Backward),Brief Visuospatial Memory Test - Revised,Hopkins Verbal Learning Test, Depression, Anxiety, Stress Scales

CONTACTS AND LOCATIONS:
Overall Officials: Paul Monagle, MD, Principal Investigator — University of Melbourne; Donald Campbell, MD, Principal Investigator — Northern Hospital
Locations (1):
- The Northern Hospital, Epping, Victoria, Australia

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the primary publication and subsequent publications(text, tables, figures, and appendices), after deidentification. Prior to releasing any data the following are required: a data access agreement must be signed between relevant parties, Study Principal Investigators must see and approve the analysis plan describing how the data will be analysed, there must be an agreement around appropriate acknowledgement and any additional costs involved must be covered. Should the Study Principal Investigators be unavailable, this role is delegated to the Murdoch Children's Research Institute. Data will only be shared with a recognised research institution which has approved the proposed analysis plan.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 6 months after primary publication of the study data for 10 years
Access Criteria: 1) Data access agreement; 2) Approval by Principal Investigators; 3) Recognised research institutions; 4) Project has received ethics approval
URL: https://www.mcri.edu.au/research/training-and-resources/launching-pad#_Data_Sharing

REFERENCES:
- [Background] Clausen TM, Sandoval DR, Spliid CB, Pihl J, Perrett HR, Painter CD, Narayanan A, Majowicz SA, Kwong EM, McVicar RN, Thacker BE, Glass CA, Yang Z, Torres JL, Golden GJ, Bartels PL, Porell RN, Garretson AF, Laubach L, Feldman J, Yin X, Pu Y, Hauser BM, Caradonna TM, Kellman BP, Martino C, Gordts PLSM, Chanda SK, Schmidt AG, Godula K, Leibel SL, Jose J, Corbett KD, Ward AB, Carlin AF, Esko JD. SARS-CoV-2 Infection Depends on Cellular Heparan Sulfate and ACE2. Cell. 2020 Nov 12;183(4):1043-1057.e15. doi: 10.1016/j.cell.2020.09.033. Epub 2020 Sep 14. PMID 32970989
- [Background] Dixon B, Smith RJ, Campbell DJ, Moran JL, Doig GS, Rechnitzer T, MacIsaac CM, Simpson N, van Haren FMP, Ghosh AN, Gupta S, Broadfield EJC, Crozier TME, French C, Santamaria JD; CHARLI Study Group. Nebulised heparin for patients with or at risk of acute respiratory distress syndrome: a multicentre, randomised, double-blind, placebo-controlled phase 3 trial. Lancet Respir Med. 2021 Apr;9(4):360-372. doi: 10.1016/S2213-2600(20)30470-7. Epub 2021 Jan 22. PMID 33493448
- [Background] van Haren FMP, Page C, Laffey JG, Artigas A, Camprubi-Rimblas M, Nunes Q, Smith R, Shute J, Carroll M, Tree J, Carroll M, Singh D, Wilkinson T, Dixon B. Nebulised heparin as a treatment for COVID-19: scientific rationale and a call for randomised evidence. Crit Care. 2020 Jul 22;24(1):454. doi: 10.1186/s13054-020-03148-2. PMID 32698853
- [Background] Conzelmann C, Muller JA, Perkhofer L, Sparrer KM, Zelikin AN, Munch J, Kleger A. Inhaled and systemic heparin as a repurposed direct antiviral drug for prevention and treatment of COVID-19. Clin Med (Lond). 2020 Nov;20(6):e218-e221. doi: 10.7861/clinmed.2020-0351. Epub 2020 Aug 30. PMID 32863274
- [Background] Mycroft-West CJ, Su D, Pagani I, Rudd TR, Elli S, Gandhi NS, Guimond SE, Miller GJ, Meneghetti MCZ, Nader HB, Li Y, Nunes QM, Procter P, Mancini N, Clementi M, Bisio A, Forsyth NR, Ferro V, Turnbull JE, Guerrini M, Fernig DG, Vicenzi E, Yates EA, Lima MA, Skidmore MA. Heparin Inhibits Cellular Invasion by SARS-CoV-2: Structural Dependence of the Interaction of the Spike S1 Receptor-Binding Domain with Heparin. Thromb Haemost. 2020 Dec;120(12):1700-1715. doi: 10.1055/s-0040-1721319. Epub 2020 Dec 23. PMID 33368089
- [Background] Tandon R, Sharp JS, Zhang F, Pomin VH, Ashpole NM, Mitra D, McCandless MG, Jin W, Liu H, Sharma P, Linhardt RJ. Effective Inhibition of SARS-CoV-2 Entry by Heparin and Enoxaparin Derivatives. J Virol. 2021 Jan 13;95(3):e01987-20. doi: 10.1128/JVI.01987-20. Print 2021 Jan 13. PMID 33173010
- [Background] Ozsoy Y, Gungor S, Cevher E. Nasal delivery of high molecular weight drugs. Molecules. 2009 Sep 23;14(9):3754-79. doi: 10.3390/molecules14093754. PMID 19783956
- [Background] Monagle K, Ryan A, Hepponstall M, Mertyn E, Monagle P, Ignjatovic V, Newall F. Inhalational use of antithrombotics in humans: Review of the literature. Thromb Res. 2015 Dec;136(6):1059-66. doi: 10.1016/j.thromres.2015.10.011. Epub 2015 Oct 9. PMID 26475409
- [Background] Figueroa JM, Lombardo ME, Dogliotti A, Flynn LP, Giugliano R, Simonelli G, Valentini R, Ramos A, Romano P, Marcote M, Michelini A, Salvado A, Sykora E, Kniz C, Kobelinsky M, Salzberg DM, Jerusalinsky D, Uchitel O. Efficacy of a Nasal Spray Containing Iota-Carrageenan in the Postexposure Prophylaxis of COVID-19 in Hospital Personnel Dedicated to Patients Care with COVID-19 Disease. Int J Gen Med. 2021 Oct 1;14:6277-6286. doi: 10.2147/IJGM.S328486. eCollection 2021. PMID 34629893
- [Background] Stelmach I, Jerzynska J, Stelmach W, Majak P, Brzozowska A, Gorski P, Kuna P. The effect of inhaled heparin on airway responsiveness to histamine and leukotriene D4. Allergy Asthma Proc. 2003 Jan-Feb;24(1):59-65. PMID 12635579
- [Background] Stelmach I, Jerzynska J, Bobrowska M, Brzozowska A, Majak P, Kuna P. [The effect of inhaled heparin on post-leukotriene bronchoconstriction in children with bronchial asthma]. Pol Merkur Lekarski. 2002 Feb;12(68):95-8. Polish. PMID 11995261
- [Background] Valencia Sanchez C, Theel E, Binnicker M, Toledano M, McKeon A. Autoimmune Encephalitis After SARS-CoV-2 Infection: Case Frequency, Findings, and Outcomes. Neurology. 2021 Dec 7;97(23):e2262-e2268. doi: 10.1212/WNL.0000000000012931. Epub 2021 Oct 11. PMID 34635560
- [Background] Misra S, Kolappa K, Prasad M, Radhakrishnan D, Thakur KT, Solomon T, Michael BD, Winkler AS, Beghi E, Guekht A, Pardo CA, Wood GK, Hsiang-Yi Chou S, Fink EL, Schmutzhard E, Kheradmand A, Hoo FK, Kumar A, Das A, Srivastava AK, Agarwal A, Dua T, Prasad K. Frequency of Neurologic Manifestations in COVID-19: A Systematic Review and Meta-analysis. Neurology. 2021 Dec 7;97(23):e2269-e2281. doi: 10.1212/WNL.0000000000012930. Epub 2021 Oct 11. PMID 34635561
- [Derived] Edwards K, Corocher T, Hersusianto Y, Campbell D, Subbarao K, Neil JA, Monagle P, Ho P. Heparin-mediated PCR interference in SARS-CoV-2 assays and subsequent reversal with heparinase I. J Virol Methods. 2024 Jun;327:114944. doi: 10.1016/j.jviromet.2024.114944. Epub 2024 Apr 20. PMID 38649069

DOCUMENTS (1):
  • Statistical Analysis Plan (2025-02-24): https://cdn.clinicaltrials.gov/large-docs/50/NCT05204550/SAP_000.pdf